## Effects of Mindfulness Training on the Psychological Well-being of Preschoolers

<u>Informed Consent Form – Parent/Guardian</u>

NCT Number: NCT05058365

Document Date: July 2021, 2021

Mindfulness Culture in Schools Initiative

Address: Room 9.30, 9/F, The Jockey Club Tower,

Centennial Campus, The University of Hong Kong,

Pokfulam Road, Hong Kong

Fax: (852) 2517 0806 (852) 3917 5176 Email: jcpanda@hku.hk Website: www.jcpanda.hk

## 樂天心澄: 靜觀校園文化計劃

Tel:

各位家長:

香港大學賽馬會「樂天心澄」 靜觀校園文化行動會於 2021-22 學年在香港基督教女青 年會戴翰芬幼兒學校試行由英國靜觀校園計劃 (Mindfulness in Schools Project, MiSP) 研發 的學前靜觀課程 - dots, 對象為 K3 學生。此項研究旨在探討靜觀課程對學前兒童身心健 康的正面影響,從而協助教育工作者提升學生的身心發展。

我們誠邀貴子弟參與是項研究計劃。參與計劃的學生會於上課時間內參加 dots 靜觀小 組,共有三十節,每節十五分鐘。每星期兩節,一共 15 周便能完成整個課程。因爲要研 究課程的成效, K3 的學生會隨機分成兩半, 一半會在上學期先上 15 週的課, 而另一半則 在下學期才上 15 週的課。在課程的前後,「樂天心澄」的研究員會從學生、老師和家長收 集數據,以評估課程的成效。數據透過遊戲、訪問和問卷來收集。

整個研究過程不會為參與者帶來任何風險。而完成此計劃有機會增加貴子弟對靜觀的 認識,從而提升他們的身心健康。在計劃完成後,我們樂意與家長、老師和同學分享整體 的研究結果。

參與此項研究純屬自願性質,所收集的資料只供研究員作研究用途,個人資料將絕對 保密。在研究過程中,參加者可以隨時停止參與而無任何不良後果。為了減省學校處理收 集回條所需的行政工作,如閣下同意貴子弟參與是項研究,則不需要任何回覆。如閣下不 希望 貴子弟參與是項研究,請於 2021 年 9 月 6 日或之前通知學校或聯絡研究員陳小姐 (3917 5176)。如閣下想知道更多有關研究參與者的權益, 請聯絡香港大學非臨床研究操 守委員會(2241 5267), 計劃編號為 EA1908007。

此致

香港基督教女青年會戴翰芬幼兒學校各家長

香港大學社會科學學院 林瑞芳教授 謹啟

主辦院校 Organised by:



揭助機構 Funded by:





Mindfulness Culture in Schools Initiative

Address: Room 9.30, 9/F, The Jockey Club Tower,

Centennial Campus, The University of Hong Kong,

Pokfulam Road, Hong Kong

Tel: (852) 3917 5176 (852) 2517 0806 Fax: Website: www.jcpanda.hk Email: jcpanda@hku.hk

Dear Parents.

## Peace and Awareness: Mindful School Culture Project

With the funding support from the Hong Kong Jockey Club Charities Trust, the Faculty of Social Sciences at the University of Hong Kong is collaborating with the school of your child to develop mindful school culture. The project aims to explore the positive effects of a mindfulness education program on students' well-being.

The program consists of 15-minute twice weekly lessons that span for fifteen weeks. Your child will be randomly assigned to the experimental group or waitlist control group. The experimental group will take the program first whereas the control group will take the program later. At the beginning and the end of the course, your child will be interviewed and will complete a computerized task. The procedure takes about 15 minutes. Parents and class teacher will also be invited to complete a short questionnaire at the beginning and the end of the course.

The research procedure has no known risk to participants. The research project can potentially enhance students' knowledge in mindfulness, which in turn enhance their well-being. It is also our pleasure to share the general results of this research with parents, teachers and students in your school once the project is completed.

Participation in the evaluation research is entirely voluntary, and all information obtained will be used for research purposes only. The data collected will only be accessed by researchers of this project. Strict confidentiality will be maintained. All the data will only be retained for 5 years after the publication of the first report. Participants will not be identified by name in any report of the completed study. They have rights to withdraw from the evaluation research at any time without negative consequences. To save the teachers' administrative work related to the collection of reply slips, no action on your part is required if you give consent for your child to participate in the study; however, if you do not wish to give consent, please make this known to the school, or contact Ms. Chan (3917 5176) before 6 September, 2021. If you want to know more about the rights of research participants, you can contact the Human Research Ethics Committee for Non-Clinical Faculties at the University of Hong Kong (2241 5267). HREC Reference Number: EA1908007.

Yours faithfully,

Lam Shui-fong

Professor

Faculty of Social Sciences The University of Hong Kong

主辦院校 Organised by:





